CLINICAL TRIAL: NCT06382116
Title: A Phase III Randomized Controlled Clinical Study Comparing BL-B01D1 With Platinum Based Chemotherapy (First-line of Systemic Treatment) in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer After EGFR-TKI Failure
Brief Title: A Study Comparing BL-B01D1 With Platinum Based Chemotherapy in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-301
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BL-B01D1 (Experimental): Participants receive BL-B01D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1
- Pemetrexed+Cisplatin or Carboplatin (Experimental): Participants receive Pemetrexed +Cisplatin or Carboplatin in the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: Pemetrexed+Cisplatin or Carboplatin

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion for a cycle of 3 weeks.
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
  Arms: BL-B01D1
Drug: Pemetrexed+Cisplatin or Carboplatin — Administration by intravenous infusion for a cycle of 3 weeks.
  Arms: Pemetrexed+Cisplatin or Carboplatin

SUMMARY:
This trial is a registered phase III, randomized, open-label, multicenter study to evaluate the efficacy and safety of BL-B01D1 in patients with locally advanced or metastatic non-squamous non-small cell lung cancer with EGFR-sensitive mutations after EGFR-TKI failure.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent and follow the requirements of the protocol;
2. Age ≥18 years old;
3. Expected survival time ≥3 months;
4. Histologically or cytologically confirmed locally advanced or metastatic non-squamous non-small cell lung cancer;
5. Documented classical EGFR mutations detected from tumor tissue or blood samples;
6. Had not received any systemic therapy other than EGFR-TKIs;
7. Radiographic disease progression documented during or after third-generation EGFR-TKI therapy for metastatic or locally advanced disease;
8. Consent to provide archival tumor tissue samples or fresh tissue samples of primary or metastatic lesions within 3 years;
9. Must have at least one measurable lesion according to RECIST v1.1 definition;
10. ECOG score 0 or 1;
11. Toxicity of previous antineoplastic therapy has returned to ≤ grade 1 defined by NCI-CTCAE v5.0;
12. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
13. The level of organ function must meet the requirements on the premise that blood transfusion is not allowed within 14 days before the screening period and no cell growth factor drugs are allowed;
14. Coagulation function: international normalized ratio (INR) ≤1.5 and activated partial thromboplastin time (APTT) ≤1.5×ULN;
15. Urine protein ≤2+ or < 1000mg/24h;
16. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before the start of treatment, serum or urine must be negative for pregnancy, and must be non-lactating; All enrolled patients (male or female) were advised to use adequate barrier contraception throughout the treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. The patient has histologic or cytologic evidence of small cell or mixed small/non-small cell component or squamous non-small cell lung cancer;
2. Chemotherapy, biological therapy, immunotherapy, etc., have been used within 4 weeks or 5 half-lives before the first dose, small molecule targeted therapy has been used within 5 days, palliative radiotherapy or anti-tumor therapy has been used within 2 weeks;
3. Previous treatment with: a. an ADC with TOPI inhibitor as toxin; b. any systemic therapy in the context of metastatic/locally advanced disease;
4. The history of severe cardiovascular and cerebrovascular diseases in the past six months prior screening;
5. Thrombotic events requiring therapeutic intervention within 6 months before screening; Infusion-related thrombosis more than 4 weeks later was excluded;
6. Complete left bundle branch block, III degree atrioventricular block, frequent and uncontrolled severe arrhythmia;
7. Other malignancies diagnosed within 3 years before randomization;
8. Hypertension poorly controlled by two antihypertensive drugs;
9. History of interstitial lung disease (ILD) requiring steroid therapy, or current ILD or grade ≥2 radiation pneumonitis;
10. Patients with poor glycemic control;
11. Complicated pulmonary diseases leading to clinically severe respiratory function impairment;
12. Patients with active central nervous system (CNS) metastases;
13. Severe infection within 4 weeks before randomization; Evidence of pulmonary infection or active pulmonary inflammation within 2 weeks before randomization;
14. Patients with massive or symptomatic effusions or poorly controlled effusions;
15. Imaging examination showed that the tumor had invaded or wrapped the abdomen, chest, neck, and large blood vessels;
16. Severe unhealed wound, ulcer, or fracture within 4 weeks before signing the informed consent;
17. Subjects with clinically significant bleeding or obvious bleeding tendency within 4 weeks before signing the informed consent;
18. Patients with inflammatory bowel disease, extensive bowel resection history, immune enteritis history, intestinal obstruction or chronic diarrhea;
19. Have a history of allergy to recombinant humanized antibodies or any of the ingredients of BL-B01D1;
20. Human immunodeficiency virus antibody positive, active hepatitis B virus infection, or hepatitis C virus infection;
21. A history of severe neurological or psychiatric illness;
22. Received other unmarketed investigational drug or treatment within 4 weeks before randomization;
23. Subjects who were scheduled to receive live vaccine or received live vaccine within 28 days before study randomization;
24. Other circumstances that were assessed by the investigator as inappropriate for participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2024-05-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  Progression-free survival (PFS) as assessed by BIRC is defined as the time between the date subjects are randomized and the first observation of disease progression (based on BICR's image-based assessment) or death.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 24 months
  Overall survival (OS) is defined as the time between the subject's randomization date and subject's death.
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective response rate (ORR) is defined as the number of CR and PR in the treatment and control groups divided by the number of that group in the full analysis set (FAS).
Disease Control Rate (DCR) | Up to approximately 24 months
  Disease Control Rate (DCR) : Percentage of all randomized subjects who rated the best overall response (BOR) as complete response (CR), partial response (PR), and disease stabilization (SD) according to RECIST 1.1 criteria.
Duration of Response (DOR) | Up to approximately 24 months
  Duration of Response (DOR) : defined as the period from the date when tumor response is first recorded to the date when objective tumor progression is first recorded or the date of death.
Treatment Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1.
Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency of anti-BL-B01D1 antibody (ADA) will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, PHD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China